CLINICAL TRIAL: NCT03109301
Title: A Phase II Trial of the Mitogen Activated Protein Kinase Kinase (MEK1/2) Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate) in Patients With Neurofibromatosis Type 1 (NF1) Mutated Gastrointestinal Stromal Tumors (GIST)
Brief Title: Mitogen Activated Protein Kinase Kinase (MEK1/2) Inhibitor Selumetinib (AZD6244 Hydrogen Sulfate) in People With Neurofibromatosis Type 1 (NF1) Mutated Gastrointestinal Stromal Tumors (GIST)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170084; 17-C-0084
Record Dates: First submitted 2017-04-11; First posted 2017-04-12 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms, Nerve Tissue; Neurofibromatosis 1; Heredodegenerative Disorders, Nervous System; Peripheral Nervous System Diseases
Keywords: Mesenchymal Neoplasm; Neurofibromatosis 1; Plexiform Neurofibromas
MeSH Terms: conditions — Neoplasms, Nerve Tissue; Neurofibromatosis 1; Heredodegenerative Disorders, Nervous System; Peripheral Nervous System Diseases; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Patients > 18 years of age
  Interventions: Drug: Selumetinib (AZD6244 hyd sulfate) 50mg/dose
- Arm 2 (Experimental): Patients < 18 years of age
  Interventions: Drug: Selumetinib (AZD6244 hyd sulfate) 25mg/m2

INTERVENTIONS:
Drug: Selumetinib (AZD6244 hyd sulfate) 50mg/dose — Selumetinib will be administered at a starting dose of 50 mg/dose orally in patients 18 years or older; drug will be given twice daily continuously in the absence of toxicity or disease progression, using 28-day cycles.
  Arms: Arm 1
Drug: Selumetinib (AZD6244 hyd sulfate) 25mg/m2 — Selumetinib will be administered at a starting dose of 25 mg/m2/dose in children < 18 years of age; drug will be given twice daily continuously in the absence of toxicity or disease progression, using 28-day cycles.
  Arms: Arm 2

SUMMARY:
Background:

Gastrointestinal stromal tumors (GIST) can cause serious medical problems. The only known treatment is surgery. But completely removing a GIST tumor with surgery is often not possible. Researchers want to see if a new drug, selumetinib, can help treat these tumors.

Objective:

To find out if selumetinib shrinks or slows the growth of GIST tumors and to see its side effects.

Eligibility:

People ages 3 and over who have one or more GIST tumors and may have neurofibromatosis type I (also called NF1). Their NF1 GIST has shown some growth or cannot be completely removed with surgery.

Design:

Participants will be screened with heart and eye tests and scans.

Participants will be told what foods and medicines they cannot take during the study. Participants will keep a diary of the medicine they take during the study.

Participants will take selumetinib capsules twice daily on an empty stomach for 28 days in a row. This is 1 cycle.

During the cycles, participants will have study visits. These may include:

Medical history

Physical exam

Blood and urine tests

Heart tests

Scans of their tumors

Eye exam

Positron emission tomography scan. They will be get radioactive glucose an IV line. They will lie quietly in a darkened room for 50-60 minutes then have the scan.

Participants will answer questions about how they are feeling.

Participants can stay in the study until they have bad side effects or their tumor grows.

After finishing treatment, participants will be watched for side effects for 30 days.

DETAILED DESCRIPTION:
BACKGROUND:

* Gastrointestinal stromal tumor (GIST) is the most common mesenchymal neoplasm of the gastrointestinal tract, and traditional cytotoxic chemotherapy is not effective. Patients with Neurofibromatosis 1 (NF1) have an increased risk of developing GIST, and surgery remains the only standard treatment option for NF1-related GIST. While the tyrosine kinase inhibitors (TKIs) imatinib and sunitinib prolong survival in patients with KIT/PDGFRA mutated GIST, they have no documented efficacy in patients with NF1 related GISTs, which lack KIT/PDGFRA mutations. Radiation therapy also seems to be ineffective. Therefore, new therapies are needed.
* Selumetinib (AZD6244 hyd sulfate), a novel orally bioavailable mitogen activated protein kinase inhibitor, is a specific inhibitor of MEK 1/2, which is currently undergoing evaluation in adults with refractory cancers, in adults and children with NF1 and plexiform neurofibromas (PN) and children with brain tumors. Evaluation of selumetinib in children and young adults with NF1 related plexiform neurofibromas (PN) has demonstrated activity with most patients demonstrating some PN shrinkage, and a partial response rate of 71%. Selumetinib has also demonstrated activity in children with NF1 and low-grade gliomas. It is thus possible that selumetinib may mediate anti-tumor effects in NF1 GIST by inhibition of downstream signaling of Ras.

OBJECTIVES:

- To estimate the response rate (radiologic response as defined by RECIST v1.1) of selumetinib in children and adults with measurable NF1-mutated GIST which is unresectable, progressive or metastatic.

ELIGIBILITY:

* Patients who are greater than or equal to 3 years of age and able to swallow capsules, with a histologically or cytologically confirmed measurable GIST without Kit or PDGFRA mutation, who have a clinical diagnosis of NF1 or a mutation of NF1 in the GIST.
* Patients tumors must demonstrate progression within the past 12 months or be metastatic; patients who do not meet this criterion will be followed, on the NF1 Natural History Study if appropriate; in the event that they demonstrate subsequent progression they may be enrolled.
* Patients must have adequate major organ function, adequate performance status, and normal LVEF by ECHO.
* No prior medical therapy is required; patients should have surgical resection if this is deemed feasible without unacceptable morbidity. Patients must meet the time requirements since prior therapy and have recovered from prior therapy toxicities.
* No prior treatment with selumetinib or another specific MEK1/2 inhibitor is permitted.

DESIGN:

* Selumetinib will be administered at a starting dose of 50 mg/dose orally in patients 18 years or older and 25 mg/m^2/dose in children < 18 years of age; drug will be given twice daily continuously in the absence of toxicity or disease progression, using 28-day cycles. The pediatric dose is the recommended phase II dose of selumetinib determined in a CTEP sponsored phase I trial of selumetinib for children and young adults with NF1 and inoperable plexiform neurofibromas, and the adult dose is equal to that used in our phase II study of adults with NF1 and inoperable PN. Adults will be allowed a one-time intrapatient dose escalation to 75mg BID provided the drug is well tolerated during the first cycle. Patients will be asked to co-enroll on POB protocol 10-C-0086: "Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies and 08-C-0079: Natural History Study and Longitudinal Assessment of Children, Adolescents, and Adults with Neurofibromatosis Type 1".
* Patients will be monitored for toxicity and response.
* Response will be assessed on a regular schedule. FDG-PET will be obtained at baseline prior to therapy, on day 11 (+/- 3 days) to assess for early FDG-PET response (optional), after 3 cycles and as clinically indicated.
* This study will use a Simon optimal two-stage phase II design with a target response rate of 25%, enrolling a minimum of 7 and a maximum of 16 evaluable patients. A maximum accrual of 20 patients may be accrued allowing for a small number (4) of inevaluable patients.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Age: greater than or equal to 3 years of age, BSA greater than or equal to 0.55 m^2, and able to swallow intact capsules.
* Diagnosis: must have either a clinical diagnosis of NF1 or a germline NF1 mutation, or in patients without the NF1 syndrome, demonstrate an NF1 mutation in the GIST verified in a CLIA certified laboratory. In patients without the NF1 syndrome, confirmation of the NF1 mutation in the GIST is required for enrollment.

  * a) For a clinical diagnosis of NF1 patients must have at least two of the diagnostic criteria for NF1 listed below

    * Six or more cafe-au-lait macules (greater or equal to 0.5cm in prepubertal subjects or greater than or equal to 1.5 cm in post pubertal subjects)
    * Freckling in axilla or groin
    * A neurofibroma or plexiform neurofibroma
    * Optic glioma
    * Two or more Lisch nodules
    * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
    * A first-degree relative with NF1
* Patients must have a histologically or cytologically confirmed measurable GIST without PDGFRA or KIT mutations. GIST may be newly diagnosed or recurrent provided that it meets criteria for progressive or metastatic disease. Metastatic disease refers to disease outside the GI tract, not simply a multifocal primary tumor. Testing performed by the Laboratory of Pathology, NCI, unless previously conducted by a CLIA/CAP external laboratory; analysis will include evaluation of 4 exons of KIT (9, 11, 13, 17) and 3 exons of PDGFRA (12, 14, 18).
* Measurable Disease:

  * Patients must have measurable GIST as defined by RECIST v 1.1 as at least one lesion not previously irradiated, that can be accurately measured at baseline greater than or equal to 10 mm in the longest diameter (except lymph nodes which must have short axis greater than or equal to 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
  * Progressive disease: GIST has demonstrated progression as defined by RECIST v1.1 within the past 12 months. Patients whose tumors do not meet this criterion, and have a diagnosis of NF1, may enroll on the NF1 Natural History study.
* Performance Status: ECOG less than or equal to 2 (Patients greater than or equal to 16 years of age must have a Karnofsky performance level of greater than or equal to 70% (or ECOG less than or equal to 2), and children less than or equal to 16 years old must have a Lansky performance of greater than or equal to 70%
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin (Hgb) greater than or equal to 9.0 g/dL
  * total bilirubin < 1.5(SqrRoot) institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 3.0 (SqrRoot) institutional upper limit of normal
  * creatinine clearance or radioisotope GFR > 60 mL/min/1.73 m^2 by either Cockcroft- Gault formula or analysis normal serum creatinine based on age described below:

    * Age (years): less than or equal to 5; Maximum Serum Creatinine (mg/dL): 0.8
    * Age (years): 5 or less or equal to 10; Maximum Serum Creatinine (mg/dL): 1.0
    * Age (years): 10 or less than or equal to 15; Maximum Serum Creatinine (mg/dL): 1.2
    * Age (years): >15; Maximum Serum Creatinine (mg/dL): 1.5
* Prior Therapy: Patients will be eligible if tumor is metastatic, unresectable, progressive, or if complete tumor resection is not considered to be feasible without substantial risk or morbidity.

  * Since there is no standard effective chemotherapy for patients with NF1 and GIST, patients may be treated on this trial without having received prior medical therapy directed at their GIST. Patients who have had prior GIST-directed surgery may enroll provided they have measurable disease.
  * Since selumetinib is not expected to cause substantial myelosuppression, there will be no limit to number of prior myelosuppressive regimen for GIST or other tumor manifestations associated with NF1.
  * Patients who have received previous investigational agents or biologic therapy, such as tipifarnib, pirfenidone, Peg-Intron, sorafenib, imatinib or other targeted therapies are eligible for enrollment. At least 4 weeks must have elapsed since receiving medical therapy directed at the PN and patients who received previous GIST-directed therapy must either demonstrate progression as defined by RECIST, or be unable to tolerate their previous therapy. Patients who received effects of all prior therapy to less than or equal to grade 1 before entering this study.
  * Cytotoxic chemotherapy last dose must have been received at least 28 days prior to enrollment, their last dose of biological therapy, immunomodulatory agents, vaccines, differentiating agents, used to treat their cancer at least 7 days prior to enrollment, their last dose of a monoclonal antibody at least 30 days prior to enrollment, and their last dose of any investigational agent at least 30 days prior

to enrollment.

* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment.
* At least 6 weeks must have elapsed prior to enrollment since the patient received any prior radiation therapy.
* At least 4 weeks must have elapsed since any surgeries, with evidence of good wound healing.

  * The effects of selumetinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 weeks after dosing with selumetinib ceases. Women of child-bearing potential must have a negative pregnancy test prior to entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform her treating physician immediately. Please note that the selumetinib

manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle.

* All patients and/or their parents or legal guardians must sign a written informed consent.
* Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
* Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g. grapefruit juice or marmalade) during the study, as these may affect selumetinib metabolism.
* Although not a requirement, participants will be asked to also participate in protocol 10-C-0086 Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies. Patients with NF1 will be asked to coenroll

on the NF1 Natural History Study and 08-C-0079: Natural History Study and Longitudinal Assessment of Children, Adolescents, and Adults with Neurofibromatosis Type 1.

EXCLUSION CRITERIA:

* Patients with evidence of another malignancy or benign tumor requiring chemotherapy or radiation therapy are excluded; however, those patients with a plexiform neurofibroma requiring treatment will be eligible as selumetinib has documented activity in plexiform neurofibromas.
* Patients with a diagnosis of NF1 and GIST who do not meet other eligibility criteria may enroll on the NF1 Natural History Study, and will be followed on this study. Should they require therapy for GIST based on evidence of progression, they may then enroll on study.
* Patients who are receiving any other investigational agents.
* Prior therapy with selumetinib or another specific MEK inhibitor is not permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib or other agents used in study.
* Previous MEK, RAS, or RAF inhibitor use.
* Patients who anticipate the need for surgical intervention within the first three cycles (3 months), as surgical intervention during the period of DLT evaluation may affect analysis of adherence and/or make the subject inevaluable.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with the following cardiac conditions are excluded:

  * Uncontrolled hypertension (Adults: blood pressure [BP] of greater than or equal to 150/95 despite medical support/management. Participants 18 years of age and younger should have a blood pressure less than or equal to 95th percentile for age, height and gender. Preexisting hypertension in adults should be controlled (either with pharmacological or nonpharmacological methods) at the time of enrollment.)
  * Acute coronary syndrome within 6 months prior to starting treatment
  * Uncontrolled angina - Canadian Cardiovascular Society grade II-IV despite medical support/management
  * Heart failure NYHA Class II or above
  * Prior or current cardiomyopathy including but not limited to the following: Known hypertrophic cardiomyopathy
  * Known arrhythmogenic right ventricular cardiomyopathy
  * Baseline left ventricular ejection fraction (LVEF) less than or equal to 55%
  * Previous moderate or severe impairment of left ventricular systolic function (LVEF less than 50% on echocardiography or equivalent on Multi-Gated Acquisition Scan [MUGA]) even if full recovery has occurred.
  * Severe valvular heart disease
  * Atrial fibrillation with a ventricular rate greater than 100 bpm on ECG at rest
* Ophthalmological conditions as follows:

  * Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion
  * Intraocular pressure (IOP) greater than 21 mmHg or uncontrolled glaucoma (irrespective of IOP).
  * Evidence of optic glioma, malignant glioma, malignant peripheral nerve sheath tumor,
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbitotemporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
  * Subjects with any other significant abnormality on ophthalmic examination (performed by an ophthalmologist) should be discussed with the Study Chair for potential eligibility.
* Inability to swallow capsules, since capsules cannot be crushed or broken.
* Patients with refractory nausea and vomiting, chronic gastrointestinal (GI) diseases (e.g., inflammatory bowel disease) or significant bowel resection that may significantly alter the absorption of study agent
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP 1A2, 2C8, 2C9, 2C19, 3A4/5 and UGT 1A1 and 1A3, P-glycoprotein, or BCRP are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* No supplementation with vitamin E is permitted because the selumetinib capsules contain vitamin E
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of selumetinib on the developing human fetus at the recommended therapeutic dose are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with selumetinib.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with selumetinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Ongoing radiation therapy, chemotherapy, hormonal therapy, immunotherapy, or biologic therapy directed at the tumor. Those patients with a plexiform neurofibroma requiring treatment will be eligible, as selumetinib has documented activity in plexiform neurofibromas.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Efficacy | End of treatment
  Estimate the response rate (radiologic response RECIST v1.1) of selumetinib in children and adults with NF1- mutated measurable gastrointestinal stromal tumor (GIST).

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)